CLINICAL TRIAL: NCT07228871
Title: Evaluation of the Effectiveness of Transcranial Magnetic Stimulation and Mirror Therapy in Hemispatial Neglect Developing After Stroke
Brief Title: The Effectiveness of Transcranial Magnetic Stimulation and Mirror Therapy in Hemispatial Neglect
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ankara Etlik City Hospital (Other Government)
Responsible Party: Principal Investigator, Ayse Naz Kalem, PM&R Specialist, Ankara Etlik City Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AEŞH-EK-2025-164
Record Dates: First submitted 2025-11-13; First posted 2025-11-14 (Actual); Last update posted 2025-11-14 (Actual); Status verified 2025-11

CONDITIONS: Hemispatial Neglect
Keywords: neglect; mirror therapy; theta burst stimulation
MeSH Terms: conditions — Perceptual Disorders | interventions — Mirror Movement Therapy; Cognitive Training

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Active cTBS + mirror therapy group (Experimental)
  Interventions: Other: Mirror Therapy; Device: cTBS; Other: Cognitive rehabilitation
- Sham cTBS + mirror therapy (Sham Comparator)
  Interventions: Other: Mirror Therapy; Other: Cognitive rehabilitation

INTERVENTIONS:
Other: Mirror Therapy — Mirror therapy will be administered 5 days a week for 2 weeks.
Device: cTBS — Patients received cTBS applied to the P3 region according to the 10/20 electroencephalogram system for 5 days a week, totalling 10 sessions over 2 weeks.
  Arms: Active cTBS + mirror therapy group
Other: Cognitive rehabilitation — Methods that facilitate adaptation in daily life activities will be taught.

SUMMARY:
The aim of this study is to evaluate the effectiveness of continuous Theta Burst Stimulation added to mirror therapy on neglect associated with stroke.

ELIGIBILITY:
Inclusion Criteria:

1. Ischemic/haemorrhagic stroke
2. Right hemisphere lesion
3. Patients with a duration of more than 7 days but less than 1 year from the date of the event
4. Aged between 18 and 75 years
5. Patients with a Mini Mental Test Score ≥ 24

Exclusion Criteria:

1. History of recurrent stroke
2. Presence of vision or hearing problems
3. Use of medication affecting cognitive function
4. History of epilepsy
5. Pregnancy or breastfeeding
6. History of malignancy
7. Pacemaker
8. Presence of metallic implants in the brain or scalp (including cochlear implant)
9. History of premorbid dementia
10. Presence of psychiatric or additional neurological disease

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Estimated)
Dates: Start 2025-10-09 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Catherine Bergego Scale | Before Treatment and 2nd week of treatment

SECONDARY OUTCOMES:
Verbal and Nonverbal Cancellation Test | Before Treatment and 2nd week of treatment
Line Bisection Test | Before Treatment and 2nd week of treatment
Barthel Index | Before Treatment and 2nd week of treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Ankara Etlik City Hospital, Ankara, Yenimahalle, Turkey (Türkiye)